CLINICAL TRIAL: NCT01809236
Title: An Open Label, Single Arm Clinical Study of Intravitreal Injection of Conbercept in Patients With Maculae Edema Secondary to Retinal Vein Occlusion (the FALCON Study)
Brief Title: Efficacy and Safety of Conbercept in Macular Edema Secondary to Retinal Vein Occlusion
Acronym: FALCON
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chengdu Kanghong Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KHSWKH902008
Record Dates: First submitted 2013-03-11; First posted 2013-03-12 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2014-03

CONDITIONS: Retinal Vein Occlusion
MeSH Terms: conditions — Retinal Vein Occlusion | interventions — KH902 fusion protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 0.5 mg Conbercept (Experimental): patients will receive monthly intravitreal injections of Conbercept to month 3 (total 3 times) and then on an as needed (PRN) dosing schedule based on the pre-specified retreatment criteria till to month 9.
  Interventions: Biological: Conbercept

INTERVENTIONS:
Biological: Conbercept — intravitreal injection of 0.5 mg Conbercept

SUMMARY:
This is a Phase II, single arm, open label clinical trial. 60 RVO patients (including 30 BRVO and 30 CRVO, respectively) are enrolled in the study. The study included a fixed treatment period (3 months) and a PRN period (6 months). In the fixed treatment period patients will receive 3 consecutive monthly intravitreal of 0.5 mg Conbercept. In the PRN period, patients are monthly visited and retreatment will be needed according to the retreatment criteria pre-specified.

ELIGIBILITY:
Inclusion Criteria:

1. Ability and willingness to provide signed Informed Consent Form.
2. Age ≥ 18, both male and female。
3. Ocular Inclusion Criterion (Study Eye):

   * Diagnosis of Foveal center-involved macular edema due to RVO (both CRVO and BRVO) within 6 months.
   * Best corrected visual acuity (BCVA) letter score in the study eye of ≤ 73（Snellen equivalents 20/40）.
   * Central retinal thickness by OCT in the study eye ≥ 320 μm.

Exclusion Criteria:

1. Brisk afferent pupillary defect.
2. History of any anti-VEGF treatment in the study and/or system within 6 months before enrollment, and/or in the fellow eye within 3 month.
3. History of intraocular and/or peri-ocular corticosteroid use in the study eye within 3 months, and/or history of use steroids systemic (p.o., i.m., i.v.) within 1 month.
4. Any active infection involving the ocular including blepharitis, infectious conjunctivitis, keratitis, scleritis, endophthalmitis in either eye.
5. Any inflammatory cells detected in the anterior chamber and/or vitreous in the study eye.
6. Presence of non-RVO disease, in the opinion of the investigator, might cause macular edema, such as AMD (wet or dry), diabetes retinopathy, uveitis etc.
7. Neovascular change in the study eye and/or neovascularization of the iris or neovascular glaucoma in study eye at baseline.
8. Patients with substantial cataract that, in the opinion of the investigator, is likely to be decreasing visual acuity by equal or more than 3 lines or medicine or surgery treatment are needed in the study eye within 4 months.
9. Patients diagnosed with systemic immune diseases and any uncontrolled clinical disease.
10. Pregnant or nursing women.
11. Patients need to exclude in the opinion of investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-05; Primary Completion 2013-11 (Actual); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in BCVA | 3-month

SECONDARY OUTCOMES:
Mean change from baseline in BCVA | baseline to 9-month
Mean change from baseline in central retinal thickness | baseline to 9-month
Mean injection times | baseline to 9-month
Mean change from baseline in Macular edema volume and other anatomical character in the study eye | baseline to 9-month
Rate of adverse event | 3-month and 9-month

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Tongren hospital affiliated to Capital Medical University, Beijing, Beijing Municipality
  - The Affiliated Eye Hospital of WMC, Wenzhou, Zhejiang